CLINICAL TRIAL: NCT05431777
Title: Retrospective, Multicenter, Observational Study to Evaluate Current Treatment Patterns and Outcomes in Japanese Patients With Locally Advanced or Metastatic Urothelial Carcinoma Treated With First-line Avelumab Maintenance
Brief Title: A Study to Learn About the Study Medicine (Avelumab) in Japanese Patients With Urothelial Carcinoma That Has Spread
Status: Completed | Type: Observational
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: B9991048
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Urothelial Carcinoma
Keywords: Retrospective; Multicenter; Observational; current treatment patterns and outcome; Avelumab; Japan; Locally advanced or metastatic urothelial carcinoma; First-line therapy
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — avelumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Japanese Patients With Locally Advanced or Metastatic Urothelial Carcinoma: Japanese Patients With Locally Advanced or Metastatic Urothelial Carcinoma who were treated with avelumab as first-line maintenance therapy
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — As provided in real world setting

SUMMARY:
The purpose of this clinical trial is to learn about the current treatment patterns, safety, and effects of the study medicine (Avelumab) for the treatment of urothelial carcinoma.

This study is seeking Japanese participants who:

* have urothelial cancer that has spread
* are treated with Avelumab for maintenance

We will study the experiences of people receiving avelumab. This helps us learn the current treatment patterns, safety, and effects of avelumab. Participants will take part in this study up to 10 months. During this time, they will have no study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with locally advanced or metastatic UC before receiving Avelumab 1L maintenance therapy.
2. Started treatment with avelumab for locally advanced or metastatic UC from 24 Feb 2021 (regulatory approval date) to 30 Nov 2021.
3. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

(1) Written consent is not required for patients who were transferred to a hospital, and registration with verbal consent is acceptable.

(2) Opt-out enrollment is allowed for patients who have already died. 4)Deceased patients are also required to meet the inclusion criteria 1)-2).

Exclusion Criteria:

There are no exclusion criteria for this study.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with locally advanced or metastatic Urothelial Carcinoma treated with first-line avelumab maintenance therapy in Japan between 24 February 2021 and 30 November 2021
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (16):
- Japan (16):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Asahi General Hospital, Asahi, Chiba
  - Kurume University Hospital, Kurume, Fukuoka
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - St. Marianna University School of Medicine, Kawasaki, Kanagawa
  - SHOWA University Fujigaoka Hospital, Yokohama, Kanagawa
  - Nara Medical University Hospital, Kashihara, Nara
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Akita University Hospital, Akita
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - University Hospital Kyoto Prefectural University of Medicine IEC, Kyoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto University Hospital, Kyoto
  - Toyama University Hospital, Toyama

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=B9991048
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled: 19-Jul-2022. Last Participant Last Visit: 16-Jan-2023
Groups:
- Avelumab in Advanced-metastatic UC: Participants diagnosed with advanced or metastatic urothelial carcinoma (UC) who were prescribed avelumab as 1L maintenance therapy between 24 February 2021 and 30 November 2021 under standard care in a real-world clinical setting in Japan.
Period: Overall Study
Arm/Group | Avelumab in Advanced-metastatic UC
Started | 79
Completed | 79
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 79
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 79
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Age of Participants at Baseline
Description: The age of participants at baseline was reported.
Time Frame: At baseline (at the initiation of avelumab maintenance therapy)
Population: Analysis set included all participants who were enrolled in the study and received maintenance avelumab treatment between 24 February 2021 and 30 November 2021, participants meeting all the inclusion criteria were analyzed.
Measure: Median (Full Range); unit: Years
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
Years | 72 [44 to 86]

2. Primary Outcome: Number of Participants With Advanced and Metastatic Urothelial Carcinoma by Sex
Description: Number of Participants With Advanced and Metastatic UC by sex was reported.
Time Frame: At baseline (at the initiation of avelumab maintenance therapy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
Participants
  Male | 60
  Female | 19

3. Primary Outcome: Number of Participants According to Location of Primary Tumor
Description: The primary tumor site is divided into the following categories: "upper urinary tract" for renal pelvis or ureter "lower urinary tract" for bladder and urethra.
Time Frame: At baseline (at the initiation of avelumab maintenance therapy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
Participants
  Bladder | 43
  Upper Tract (renal pelvis or ureter) | 36

4. Primary Outcome: Number of Participants With Presence of Urothelial Carcinoma Subtype
Description: The subtype of urothelial carcinoma included micropapillary, microcystic, nested, lymphoepithelioma-like, plasmacytoid, sarcomatoid, giant cell, poorly differentiated, lipid rich, clear cell. number of participants with presence of UC subtype was reported.
Time Frame: At baseline (at the initiation of avelumab maintenance therapy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
Participants
  No | 33
  Yes | 13
  Unknown | 20
  Not reported | 13

5. Primary Outcome: Number of Participants With Metastatic Sites at Start of First Line Chemotherapy
Description: Number of participants with metastatic sites at start of First Line Chemotherapy was reported.
Time Frame: At baseline (at the initiation of avelumab maintenance therapy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
Participants
  Single | 18
  Multiple | 34
  None | 25
  Unknown | 2

6. Primary Outcome: Number of Participants With Eastern Cooperative Oncology Group Performance Status (ECOG PS) at Start of First Line Chemotherapy
Description: ECOG PS measured on-therapy (time between first dose and last dose date) assessed participant's performance status on 5 point scale: 0 is equal to (=) fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (greater than [>] 50% of waking hours [hrs]), capable of all self care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hrs; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=dead.
Time Frame: At the initiation of first line chemotherapy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
Participants
  0 | 56
  1 | 19
  2 | 3
  3 | 1
  4 | 0

7. Primary Outcome: Number of Participants Who Received First Line (IL) Chemotherapy Regimens
Description: Chemotherapies were categorized as: 1.Gemcitabine + Cisplatin 2. Gemcitabine + Carboplatin 3. Dose-dense methotrexate, vinblastine, doxorubicin, cisplatin 4. Other.
Time Frame: At baseline (at the initiation of avelumab maintenance therapy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
Participants
  Gemcitabine + Cisplatin | 50
  Gemcitabine + Carboplatin | 24
  Dose-dense methotrexate, vinblastine, doxorubicin, cisplatin | 2
  Other | 3

8. Primary Outcome: Number of First Line Chemotherapy Cycles
Description: Number of Firstline Chemotherapy Cycles in participants at baseline was reported.
Time Frame: At baseline (at the initiation of avelumab maintenance therapy)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: cycles
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
cycles | 4 [4 to 6]

9. Primary Outcome: Number of Participants With Best Response to First Line Chemotherapy According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator
Description: Determination of the best overall response to first-line chemotherapy is categorized as following: "Objective response" when "Complete Response" or "Partial Response." "Non-objective response" when "Stable Disease" of "Progressive Disease"
Time Frame: At baseline (at the initiation of avelumab maintenance therapy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
Participants
  Complete Response | 8
  Partial Response | 46
  Stable Disease | 25
  Progressive Disease | 0

10. Primary Outcome: Number of Participants With Presence or Absence of Variant Histology
Description: Number of participants with presence or absence of variant histology was reported.
Time Frame: At baseline (at the initiation of avelumab maintenance therapy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
Participants
  Presence | 13
  Absence | 33
  Unknown | 20
  Not Reported | 13

11. Primary Outcome: Treatment-Free Interval
Description: Treatment free-interval is defined as the time from the end date of first-line chemotherapy to the start date of avelumab administration. Treatment-free interval divided into the following categories. <4 weeks/4 to 10 weeks/>10 weeks.
Time Frame: At baseline (at the initiation of avelumab maintenance therapy)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
days | 34 [12 to 371]

12. Primary Outcome: Percentage of Participants With Second-Line Treatment Regimen
Description: Second-Line Therapies were categorized as: 1. Platinum Chemotherapy, 2. Enfortumab Vedotin, Gem, Gemcitabine, 3.immune checkpoint inhibitor.
Time Frame: At baseline (at the initiation of avelumab maintenance therapy)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
percentage of participants
  Platinum Chemotherapy | 51.4
  Enfortumab Vedotin | 35.1
  Immune Checkpoint Inhibitor | 8.1
  Others | 5.4

13. Secondary Outcome: Time to Failure (TTF) of Avelumab
Description: TTF was defined as the time from start of avelumab maintenance therapy to the date of end of treatment due to any cause including death. If there is no record of the end of treatment, it be discontinued on the last visit date during the study period.
Time Frame: Time from start of avelumab maintenance therapy to the date of end of treatment due to any cause including death, assessed up to 5.9 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
months | 4.57 [3.30 to 6.37]

14. Secondary Outcome: Real-World Progression-Free Survival (Rw-PFS)
Description: rwPFS is defined as: The time from start of avelumab maintenance therapy to date of first disease progression (as clinically assessed by local investigator based on radiology, laboratory evidence, pathology, or other assessments) or death due to any cause, whichever occurred first. If there were no clinical records of death or disease progression, they will be censored at the date of initiation of the next line of therapy for the participants undertaking 2 or more lines of therapy (subsequent therapy after avelumab maintenance therapy) based on the record, or at their last visit date during the study period for the participants undertaking only 1 line of therapy (only avelumab maintenance therapy) based on the record.
Time Frame: From index date up to 30 Jun 2022, where index date was date of first prescription for avelumab between 24 February 2021 and 30 November 2021 (maximum observation period was of 16 months approximately)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
Months | 6.10 [3.63 to 9.67]

15. Secondary Outcome: Overall Response Rate (ORR)
Description: The Best ORR was defined as the percentage of participants having achieved complete response (CR) or partial response (PR) according to RECIST version 1.1 as determined by the IRC. CR: defined as disappearance of all target and all non-target lesions and no new lesions. PR: defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters, no progression of non-target lesions and no new lesions.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 79
percentage of participants | 31.6 [21.6 to 43.1]

16. Secondary Outcome: Real-World Progression-Free Survival (Rw-PFS) From Chemotherapy (rwPFS-c）
Description: rwPFS-c is defined as the following: The time from start of first-line Chemotherapy to date of first disease progression (as clinically assessed by local investigator based on radiology, laboratory evidence, pathology, or other assessments) or death due to any cause during avelumab treatment, whichever occurred first. If there were no clinical records of death or disease progression, they will be censored at the date of initiation of the next line of therapy for the participants undertaking 2 or more lines of therapy (subsequent therapy after avelumab maintenance therapy) based on the record, or at their last visit date during the study period for the participants undertaking only 1 line of therapy (only avelumab maintenance therapy) based on the record.
Time Frame: as for outcome 13
Population: According to protocol, only participants whose best overall response to chemotherapy was assessed as CR, PR,orSD received avelumab treatment,and their PFS was evaluated.However,for participants whose best overall response to chemotherapy was assessed as Progressive Disease,data on subsequent treatment regimens and PFS were not collected. Due to this selective data collection,the data would not be representative of the rwPFS-c for the patient population.For these reasons data was not collected.
Arm/Group | Avelumab in Advanced-metastatic UC
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Due to non-interventional nature of study, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not meet, hence adverse events were not observed.
Arm/Group | Avelumab in Advanced-metastatic UC
All-Cause Mortality (participants affected / at risk) | 0/79
Serious Adverse Events (participants affected / at risk) | 0/79
Other Adverse Events (participants affected / at risk) | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT05431777/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT05431777/SAP_001.pdf